CLINICAL TRIAL: NCT06801535
Title: Efficacy of 3D-Printed Mouth Splints in the Management of Microstomia in Burn Patients
Brief Title: Efficacy of 3D-Printed Mouth Splints
Acronym: 3DMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00124137
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Microstomia
Keywords: cleft lip and palate; craniocarpotarsal dysplasia; dental hygiene
MeSH Terms: conditions — Microstomia; Cleft Lip; Freeman-Sheldon syndrome | interventions — Splints

STUDY DESIGN:
Intervention Model Description: Assess the impact of the 3D-printed mouth splint on oral aperture measurements over a 3-month period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Assess the impact of the 3D-printed mouth splint on oral aperture measurements over a 3-month period.
  Interventions: Device: Splint

INTERVENTIONS:
Device: Splint — Patients will use the splint at home 3 times daily for 10 minutes per session for 3 months total.

SUMMARY:
The study will investigate the effectiveness of a 3D-printed mouth splint designed to increase dimensions of oral aperture and reduce disability associated with mouth contractures. The validated Mouth Impairment and Disability Assessment (MIDA) survey will be used to objectively measure patient progress in functionality and quality of life.

DETAILED DESCRIPTION:
Microstomia, or reduced oral aperture, is a debilitating condition that can arise after burn injuries, particularly to the face. This condition severely impacts oral hygiene, nutrition, speech, and overall quality of life. Current management strategies often rely on therapy, surgical intervention, and splinting to improve mouth opening and functionality. However, there is a lack of accessibility to good mouth splinting devices. 3D-printed, dynamic splints offer may offer a superior and cost-effective solution that can be tailored to the patient's anatomy while allowing for at-home treatment. Sizing can also be adjusted to fit essentially any aperture since, including pediatrics. This device is intended for use at home, supported by teaching and follow-up provided by occupational therapists (OTs).

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years to 99 years of age with documented microstomia following burn injuries.
* Ability to comply with prescribed home exercises and follow-up visits.

Exclusion Criteria:

* Cognitive or physical inability to perform the prescribed exercises.
* Inability of a caretaker to be able to deliver therapy daily.
* Concomitant conditions that may significantly affect oral aperture (e.g., temporomandibular joint (TMJ) disorders).

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Aperture measurements | Baseline to Month 3
  Difference in measurements of oral aperture from Baseline visit to Final visit will be reported - Oral aperture measurements taken with calipers

SECONDARY OUTCOMES:
Change in Mouth Impairment and Disability Assessment (MIDA) Scores | Baseline to Month 3
  The mouth impairment and disability assessment (MIDA) has a 28 item self-report portion, divided into four subscales, completed by the patient and an impairment-based section completed by the burn therapist. The Mouth Impairment and Disability Assessment (MIDA) scale typically ranges from a low score indicating minimal impairment to a high score representing significant disability, with the exact range depending on the specific version of the scale and how individual items are scored; however, most versions will have a total score that can be interpreted within a broader range of severity, with higher scores signifying greater impairment. This assessment is scored from 0 to 64. Zero is equivalent to no difficulty and 64 would indicate the highest level of difficulty.
Change in Patient Satisfaction Scores | Baseline to Month 3
  Total patient satisfaction scored on survey at weekly visits to be reported from 0 to 23. 0 equivalent to no satisfaction and 23 is the highest level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Runyan, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Couture MA, Calva V, de Oliveira A, LaSalle L, Forget N, Nedelec B. Development and clinimetric evaluation of the mouth impairment and disability assessment (MIDA). Burns. 2018 Jun;44(4):980-994. doi: 10.1016/j.burns.2017.10.024. Epub 2018 Feb 7. PMID 29428487